CLINICAL TRIAL: NCT01025570
Title: A Study Evaluating Safety and Efficacy of Gemcitabine Plus Bosutinib for Patients With Resected Pancreatic Adenocarcinoma
Brief Title: A Study Evaluating Gemcitabine Plus Bosutinib for Patients With Resected Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09456; 10-00560 (Other: UCSF CHR-approval number)
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; pancreatic; bosutinib; SKI-606; gemcitabine; gemzar; Patients with resected pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gem/Bos (Experimental): Gemcitabine 1000 mg/m2, D1,8,15 of each cycle
  Bostutinib 400 mg daily concurrently with Gemcitabine
  Interventions: Drug: Gemcitabine, Bosutinib

INTERVENTIONS:
Drug: Gemcitabine, Bosutinib — Gemcitabine, 1000 mg/m2 on D1,8,15 over 30 mins standard infusion rate Bosutinib 400 mg, oral, once daily

SUMMARY:
The purpose of this study is to find out the effects, good and/or bad, of the combination of two drugs, gemcitabine and bosutinib, in patients with resected pancreatic cancer and whether this combination can prevent pancreatic cancer from coming back.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the pancreas.
* Complete resection by standard pancreaticoduodenectomy (for tumors of the pancreatic head) or distal pancreatectomy (for tumors of the pancreatic tail). Positive microscopic margins are allowable.
* No measurable disease.
* ECOG performance status 0 - 1.
* ≥ 18 years of age.
* Ability to start adjuvant therapy within 8 weeks after pancreatic cancer surgery (but no sooner than 3 weeks).
* CA 19-9 ≤ 2.5 times the upper limit of normal.
* ANC (absolute neutrophil count) ≥ 1500/μL
* Hemoglobin ≥ 9 gm/dL (may be transfused or may receive epoetin alfa to maintain this level)
* Platelet count ≥ 100,000/μL
* INR ≤ 1.5 (except those subjects who are receiving full-dose warfarin)
* Total bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times the upper limit of normal
* Serum creatinine ≤ 2.0
* Negative pregnancy test for women of childbearing potential (serum or urine beta-HCG).
* All patients must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.
* Women or men of reproductive potential must agree to use an effective contraceptive method during treatment and for 6 months afterwards.
* At least one paraffin block from patient's pancreatic cancer surgery must be available for analysis (does not necessarily need to be received by the start of study treatment).

Exclusion Criteria:

* Any prior systemic or investigational therapy for pancreatic cancer.
* Grossly positive surgical margins.
* Any of the following post-operative complications: wound dehiscence or infection, intraabdominal abscess, pancreatic or biliary leak or fistula.
* History of major psychiatric disorder or other chronic medical illness that, in the opinion of the treating physician, contraindicates the use of the investigational drugs in this protocol or that might render the subject at high risk of treatment related complications.
* Serious active ongoing infection, including any requiring parenteral antibiotics.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse.
* Pregnancy (positive pregnancy test) or lactation.
* Known central nervous system disease.
* Inability to swallow pills/tolerate oral intake.
* Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of using the combination of gemcitabine and bosutinib in the postoperative adjuvant treatment of patients with completely resected pancreatic cancer. | 8 weeks after the 6th patient is enrolled
To estimate the median disease-free survival rate of patients with completely resected pancreatic cancer treated with this combination | 2 years after last patient is enrolled

SECONDARY OUTCOMES:
To determine the overall survival rates of patients with completely resected pancreatic cancer when treated postoperatively with the combination of gemcitabine and bosutinib | 2 years after last patient is enrolled
To estimate both disease-free and overall survival at one and two years of patients with completely resected pancreatic cancer treated with this combination | 2 years after last patient is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Ko, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah